CLINICAL TRIAL: NCT00491608
Title: A Phase 3b, Open-Label, Single-Group Immunogenicity and Safety Study of Topical Recombinant Thrombin (rThrombin) in Surgical Hemostasis
Brief Title: Immunogenicity and Safety Study of Topical Recombinant Thrombin in Surgical Hemostasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZymoGenetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 499F04
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Results first posted 2012-01-12 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Spinal Surgery; Vascular Surgery
Keywords: Phase 3b; rThrombin; spine surgery; vascular surgery; hemostasis; immunogenicity; safety
MeSH Terms: interventions — recombinant human thrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): rThrombin
  Interventions: Biological: rThrombin

INTERVENTIONS:
Biological: rThrombin — 1000 U/mL applied directly or in combination with absorbable gelatin sponge or powder

SUMMARY:
The purpose of this study is to evaluate the safety and immune system response to recombinant thrombin when used to control bleeding in spinal and vascular surgery.

DETAILED DESCRIPTION:
This is a Phase 3b, open-label, single-group, multisite safety and immunogenicity study of recombinant thrombin (rThrombin) in participants who are at least 18 years of age and undergoing spinal or vascular surgery. Eligible participants will receive topical rThrombin during surgery and complete a 1-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Currently undergoing cervical, thoracic, or lumbar discectomy; corpectomy, laminectomy, lateral or interbody fusion, including both anterior and posterior approaches (not including minimally invasive procedures; arterial reconstruction; peripheral artery bypass (PAB) grafting; or arteriovenous (AV) vascular access procedures
* History of surgery with high likelihood of exposure to bovine thrombin within the past 3 years. Prior surgery must have been 1 of the following open procedures: open procedures involving the spine or cranium, PAB grafting, AV vascular access procedures, autologous skin grafting, or other surgical procedure accompanied by documented treatment with bovine thrombin
* Age of 18 years or younger at time of informed consent
* If female and of child-bearing potential: Negative pregnancy test result within 14 days prior to treatment
* Use of a medically accepted form of contraception from the time of informed consent to completion of all follow-up study visits, if sexually active male or a sexually active female of childbearing potential
* Signed IRB/independent ethics committee-approved informed consent document

Exclusion Criteria:

* Currently undergoing procedures requiring cardiopulmonary bypass or involving the aortic arch
* Known hypersensitivity to rThrombin or any of its components
* Presence of medical, social, or psychosocial factors that, in the opinion of the investigator, could impact safety or compliance with study procedures
* Breastfeeding
* Receipt of treatment with any experimental agent within 30 days of study enrollment or treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Alexander, MD, CPI, Study Director — ZymoGenetics
Locations (1):
- Huntington Memorial Hospital, Pasadena, California, United States

REFERENCES:
- [Derived] Randleman CD Jr, Singla NK, Renkens KL, Souza S, Pribble JP, Alexander WA. Persistence of antibodies to the topical hemostat bovine thrombin. J Am Coll Surg. 2010 Dec;211(6):798-803. doi: 10.1016/j.jamcollsurg.2010.07.023. Epub 2010 Oct 25. PMID 20980172
- [Derived] Singla NK, Ballard JL, Moneta G, Randleman CD Jr, Renkens KL, Alexander WA. A phase 3b, open-label, single-group immunogenicity and safety study of topical recombinant thrombin in surgical hemostasis. J Am Coll Surg. 2009 Jul;209(1):68-74. doi: 10.1016/j.jamcollsurg.2009.03.016. Epub 2009 May 28. PMID 19651065

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 234 participants enrolled, 209 received study drug. Of those who received study drug, 200 had both baseline and post-baseline immunogenicity evaluations.
Groups:
- rThrombin, 1000 IU/mL: Participants received at least 1 application of recombinant thrombin (rThrombin), 1000 IU/mL, during a single surgical procedure. rThrombin was applied, per investigator judgment and standard clinical practice, directly or in combination with an absorbable gelatin sponge or powder.
Period: Overall Study
Arm/Group | rThrombin, 1000 IU/mL
Started | 209 (Participants who received treatment)
Completed | 206
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- rThrombin: Participants who received at least 1 application of rThrombin during spinal or vascular surgery (arterial reconstruction or PAB,or AV vascular access procedure and had seronegative baseline rThrombin antibody status
Arm/Group | rThrombin
Number analyzed (Participants) | 209
Age, Customized [Median (Full Range); unit: Years]
  Overall (All status) | 64 [30 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 110
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 25
  Asian | 2
  Black or African American | 22
  White | 160

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anti-recombinant Thrombin (rThrombin) Product Antibodies at Day 29 in Participants With and Without Anti-bovine Thrombin Product Antibodies at Baseline
Description: Seropositive=with specific anti-bovine thrombin product antibodies; seronegative=without specific anti-bovine thrombin product antibodies.
Time Frame: At Day 29
Population: Participants who received treatment with rThrombin and had results from both baseline and post-baseline antibody assessments
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 200
Participants
  Seropositive at baseline (n=31) | 0
  Seronegative at baseline (n=169) | 0
  Total (all participants) | 0

2. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events, Treatment-related Adverse Events (AEs), and Treatment-emergent AEs
Description: AE=a new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may or may not have a causal relationship with treatment. SAE=an unfavorable medical event that results in death, persistent or significant incapacity, or drug dependency or abuse; is life-threatening, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=possibly, probably, or certainly related to study drug. Treatment-emergent=onset on or after treatment start. Grade (Gr) 1=mild, Gr 2=moderate, Gr 3=severe, Gr 4=life threatening/disabling, Gr 5=death.
Time Frame: Day 1 (surgery) to Day 29 (end of study), continuously
Population: All participants who received at least 1 application of rThrombin during surgery.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 209
Participants
  Deaths | 2
  Serious adverse events | 47
  Treatment-related adverse events (AEs) | 4
  Treatment-emergent AEs ≥ Grade 3 | 76
  AEs leading to discontinuation | 0

3. Secondary Outcome: Number of Participants With Abnormal Hematology Laboratory Results of Common Terminology Criteria (CTC) Grade 2 or Higher at Baseline and Day 29
Description: Hemoglobin, low (g/L): Grade 2=<100 Grade 3=<80; Grade 4=<65. Platelets, low: Grade 2=<75*10^9/L; Grade 3=<50*10^9/L; Grade 4=<25*10^9/L. Leukocytes, low: Grade 2=<3.0-2.0*10^9/L; Grade 3=<2.0-1.0*10^9/L; Grade 4=<1.0*10^9/L. Lymphocytes, low: Grade 2=<0.8*10^9/L; Grade 3=<0.5*10^9/L; Grade 4=<0.2*10^9/L. Neutrophils, low: Grade 2=<1.5*10^9/L; Grade 3=<1.0*10^9/L; Grade 4=<0.5*10^9/L. Changes in hematocrit values observed were not graded for severity.
Time Frame: Baseline and Day 29 (end of study)
Population: All participants who who received at least 1 application of rThrombin during surgery and had laboratory test results available for baseline and Day 29 visits.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 209
Participants
  Hemoglobin, low: Baseline, Grade 2 (n=199) | 13
  Hemoglobin, low: Day 29, Grade 2 (n=196) | 12
  Hemoglobin, low: Baseline, Grade 3 (n=199) | 3
  Hemoglobin, low: Day 29, Grade 3 (n=196) | 0
  Hemoglobin, low: Baseline, Grade 4 (n=199) | 0
  Hemoglobin, low: Day 29, Grade 4 (n=196) | 0
  Platelets, low: Baseline Grade 2 (n=196) | 0
  Platelets, low: Day 29, Grade 2 (n=194) | 1
  Platelets, low: Baseline, Grade 3 (n=196) | 1
  Platelets, low: Day 29, Grade 3 (n=194) | 0
  Platelets, low: Baseline, Grade 4 (n=196) | 0
  Platelets, low: Day 29, Grade 4 (n=194) | 0
  Leukocytes, low: Baseline, Grade 2 (n=199) | 1
  Leukocytes, low: Day 29, Grade 2 (n=196) | 0
  Leukocytes, low: Baseline, Grade 3 (n=199) | 0
  Leukocytes, low: Day 29, Grade 3 (n=196) | 0
  Leukocytes, low: Baseline, Grade 4 (n=199) | 0
  Leukocytes, low: Day 29, Grade 4 (n=196) | 0
  Lymphocytes, low: Baseline, Grade 2 (n=199) | 6
  Lymphocytes, low: Day 29, Grade 2 (n=196) | 6
  Lymphocytes, low: Baseline, Grade 3 (n=199) | 0
  Lymphocytes, low: Day 29, Grade 3 (n=196) | 2
  Lymphocytes, low: Baseline, Grade 4 (n=199) | 0
  Lymphocytes, low: Day 29, Grade 4 (n=196) | 0
  Neutrophils, low: Baseline, Grade 2 (n=199) | 1
  Neutrophils, low: Day 29, Grade 2 (n=196) | 1
  Neutrophils, low: Baseline, Grade 3 (n=199) | 1
  Neutrophils, low: Day 29, Grade 3 (n=196) | 0
  Neutrophils, low: Baseline, Grade 4 (n=199) | 0
  Neutrophils, low: Day 29, Grade 4 (n=196) | 0

4. Secondary Outcome: Number of Participants With Elevations in Coagulation Parameters of CTC Grade 3 or Higher at Baseline and Day 29
Description: Activated partial thromboplastin time (aPTT) elevations: Grade 3=>2*upper limit of normal (ULN). International normalized ratio(INR)elevations: Grade 3=>2*ULN. Changes in prothrombin time were not graded for toxicity. n=Number of participants with assessments available at that visit.
Time Frame: Baseline and Day 29 (end of study)
Population: All participants who received at least 1 application of rThrombin during surgery and had laboratory test results available for assessment.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 209
Participants
  aPTT: Baseline, Grade 3 (n=197) | 6
  aPTT: Day 29: Grade 3 (n=199) | 7
  INR: Baseline, Grade 3 (n=197) | 1
  INR: Day 29: Grade 3 (n=198) | 1

5. Secondary Outcome: Number of Participants With Abnormal Laboratory Results in Median Levels of Immunoglobulin A, G, and M at Baseline or Day 29
Description: Abnormal laboratory findings were recorded as AEs when the investigator considered them to be clinically significant (eg, an unusual result for the surgical population or for an individual participant) or when they were associated with symptoms or required treatment or a change in patient management.
Time Frame: Baseline and Day 29 (end of study)
Population: All participants who received rThrombin and had both baseline and postbaseline antibody assessments available.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 200
Participants | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Changes in Mean Values for Vital Signs (Temperature, Systolic Blood Pressure, Diastolic Blood Pressure, Respiration Rate, Heart Rate) at Baseline and Day 29
Description: Laboratory findings considered clinically significant by investigator when associated with symptoms, required specific treatment, or required a change in participant management. Clinically significant changes in vital signs were reported as adverse events.
Time Frame: Baseline and Day 29 (end of study)
Population: All participants who received at least 1 application of rThrombin during surgery.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 209
Participants | 0

ADVERSE EVENTS:
Arm/Group | rThrombin, 1000 IU/mL
Serious Adverse Events (participants affected / at risk) | 47/209
Other Adverse Events (participants affected / at risk) | 197/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rThrombin, 1000 IU/mL (N=209)
Atrial fibrillation (Cardiac disorders) | 3
Deep vein thrombosis (Vascular disorders) | 3
Hyperkaleamia (Metabolism and nutrition disorders) | 3
Myocardial infarction (Cardiac disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Wound secretion (Injury, poisoning and procedural complications) | 3
Cardiac failure congestive (Cardiac disorders) | 2
Hematoma (Vascular disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Postoperative wound infection (Infections and infestations) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 2
Abdominal wall hematoma (Gastrointestinal disorders) | 1
Acute polyneuropathy (Nervous system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Arteriovenous fistual occlusion (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1
Arteriovenous graft site haematoma (Vascular disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bacteremia (Infections and infestations) | 1
Cardiac arrest (Cardiac disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Gastroenteritis viral (Infections and infestations) | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1
Hemorrhage (Vascular disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Impaired healing (General disorders) | 1
Incision site infection (Infections and infestations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1
Renal failure acute (Renal and urinary disorders) | 1
Sedation (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 1
Spinal cord injury lumbar (Injury, poisoning and procedural complications) | 1
Steal syndrome (Vascular disorders) | 1
Stent-graft endoleak (Injury, poisoning and procedural complications) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Syncope (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 1
Transient ischemic attack (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Wound infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rThrombin, 1000 IU/mL (N=209)
Nausea (Gastrointestinal disorders) | 56
Constipation (Gastrointestinal disorders) | 42
Vomiting (Gastrointestinal disorders) | 19
Pyrexia (General disorders) | 20
Edema peripheral (General disorders) | 16
Incision site pain (Injury, poisoning and procedural complications) | 94
Procedural pain (Injury, poisoning and procedural complications) | 82
Wound secretion (Injury, poisoning and procedural complications) | 13
Hypokalemia (Metabolism and nutrition disorders) | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17
Headache (Nervous system disorders) | 17
Insomnia (Psychiatric disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 15
Hypotension (Vascular disorders) | 23
Anemia (Blood and lymphatic system disorders) | 35
Sinus tachycardia (Cardiac disorders) | 12
Tachycardia (Cardiac disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ZymoGenetics (ZG) agreements vary by trial, but each states that presentation/publication (p/p) cannot disclose Confidential Information (CI), excluding trial results; p/p may not begin until the earlier of 18 months after study end, ZG/lead investigator publishes, or ZG notification that multicenter publication is not planned; ZG has specified time for draft review before submission/presentation and may delay or modify content, require CI removal, and delay p/p for patent application filing.